CLINICAL TRIAL: NCT06566404
Title: Gene Expression Profiles and ctDNA for Risk Stratification in Patients With Melanoma Eligible for Lymph Node Sentinel Biopsy (CORRESPOND): an Observational Prospective Study.
Brief Title: Gene Expression Profiles and ctDNA for Risk Stratification in Patients With Melanoma
Acronym: CORRESPOND
Status: Not yet recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: L2-095
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Melanoma
Keywords: Melanoma; MerlinTM; ctDNA; sentinel lymph node status
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All included patients will undergo blood collection for liquid biopsy and biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at assessing the role of MerlinTM and ctDNA in predicting the nodal status in patients with >pT3b melanoma, therefore candidate for adjuvant therapy regardless of sentinel lymph node status.

DETAILED DESCRIPTION:
Cutaneous melanoma is a malignancy arising from melanocytes of the skin. Incidence rates are rising, particularly in White populations.

For patients with clinically node-negative (cN0) disease, sentinel lymph node biopsy (SLNB) is indicated for all patients with a melanoma of thickness of 0.8 mm or more (>pT1b) to stratify the prognosis and guarantee access to systemic adjuvant treatments.

Indeed, adjuvant immune checkpoint inhibitors or anti-proto-oncogene B-Raf (anti- BRAF) / Mitogen-activated protein kinase kinase (MEK) targeted agents were first demonstrated to improve clinical outcomes in patients with nodal involvement (stage III melanoma). Subsequently, immune-checkpoint inhibitors demonstrated a benefit in terms of disease-free survival also in patients with stage IIB and IIC melanoma, i.e., with melanoma of thickness of 2 mm or more (>pT3b). As a consequence, in this subgroup of patients, SLNB has lost its therapeutical implications and maintains only a role for prognostication, i.e., in the distinction between stages IIB-IIC (SLNB-negative; 71% of cases) and stage III (SLNB-positive; 29% of cases).

However, SLNB can be complicated by seroma, bleeding, wound infection, nerve damage, and even low rates of lymph edema have been reported. Moreover, depending on the country and healthcare system, it is a costly procedure for patients and society. According to an idea of professor Umberto Veronesi, Gentilini et al. demonstrated that the omission of SLNB in patients with cT1N0M0 breast cancer has not an impact on distant disease-free survival at 5 years (SOUND trial). Novel prognostic biomarkers for melanoma can substitute the SLNB role in prognostication and eventually lead to SLNB de-escalation.

Gene expression profiles (GEPs) and circulating tumor DNA (ctDNA) represents promising methods to assess tumor burden and tumor invasiveness, thus stratifying the prognosis.

ctDNA demonstrated to predict recurrence in patients with resected stage II-III melanoma, with a sensitivity and a specificity of 11-80% and 55-100%, according to the method (tumor-informed vs. tumor-naive), the techniques (digital droplet PRC [ddPCR] or others), the approach (single time point vs. dynamic assessment). In patients with non-resected stage II-III melanoma, the ctDNA-positivity rate is 35-37%. However, no data about pre-operative ctDNA as a predictor of SLNB status is available.

GEPs, alone or combined with clinicopathological features (CP-GEP), demonstrated to predict outcomes in patients with non-metastatic melanoma. In particular, MerlinTM assay is a CP-GEP model, developed by logistic regression modeling, which combines clinicopathologic factors (age and Breslow thickness) with the gene expression profiling component of 8 specific genes involved in cancer metastasis and melanosome biogenesis. It identifies patients at high or low risk of nodal metastasis. However, most patients included in studies validating this assay had a pathologic tumore stage 1-2 (pT1-2) melanoma; in patients with pathologic tumore stage 3 (pT3) melanoma this assay is characterized by high sensitivity but low specificity, and a negative predictive value of 75%.

The combination of CP-GEP and ctDNA may improve the prognostication and the prediction of SLNB status in patients with a >pT3b melanoma (candidate to adjuvant therapy regardless of nodal status), eventually leading to the de-escalation of SLNB. Indeed, in this population, in case of concordance between biomarker-positivity and SLNB status, SLNB can be definitively omitted, without missing any information.

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged at least 18 years;
* histologically documented melanoma;
* thickness > 2 mm (>pT3b);
* clinical node-negative (cN0) and non-metastatic (cM0) disease at ultrasound (US) and computed tomography (CT) or positron emission tomography (PET) scan;
* known BRAF, N-ras proto-oncogene (NRAS) and tyrosine-protein kinase (c-KIT) mutational status;
* candidate to SLNB;
* consent for the provision of plasma samples for ctDNA analysis and tissue samples (at a central laboratory).

Exclusion Criteria:

* SLNB performed;
* receipt of neoadjuvant therapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CORRESPOND is a prospective, longitudinal, observational, non-interventional, translational clinical study enrolling patients with non-metastatic node-negative melanoma.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Model Performance | 36 months
  to compare the performance of the clinicopathologic model and the clinicopathologic model including ctDNA and MerlinTM in predicting SLNB-positivity in terms of area under receiver operating characteristic curve (AUC)

SECONDARY OUTCOMES:
the estimation of the correlation between ctDNA-positivity and SLNB-positivity | 36 months
  to assess the role of ctDNA-detected mutations in predicting the SLNB status
The estimation of the correlation between MerlinTM/ctDNA-positivity and SLNB-positivity | 36 months
  To assess the role of MerlinTM and ctDNA in predicting micro- or macro- SLNB involvement (micrometastasis [TNM pathologic stage N1a (pN1a) or N2a (pN2a)] vs. macrometastasis [TNM pathologic stage N1b (pN1b) or N2b (pN2b]).

OTHER OUTCOMES:
The threshold of ctDNA Variant Allele Frequency (VAF) | 36 months
  The threshold of ctDNA VAF corresponding to nodal status with the highest accuracy (ROC analysis)
The estimation of the correlation between ctDNA-positivity and SLNB-positivity | 36 months
  The estimation of the correlation between ctDNA-positivity and SLNB-positivity according to molecular alterations detected from the ctDNA
The estimation of the correlation between features | 36 months
  The estimation of the correlation between features identified by digital pathology tecniques and SLNB-positivity

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Pennacchioli, MD, Principal Investigator — Istituto Europeo di Oncologia

REFERENCES:
- [Background] Long GV, Swetter SM, Menzies AM, Gershenwald JE, Scolyer RA. Cutaneous melanoma. Lancet. 2023 Aug 5;402(10400):485-502. doi: 10.1016/S0140-6736(23)00821-8. Epub 2023 Jul 24. PMID 37499671
- [Background] Gentilini OD, Botteri E, Sangalli C, Galimberti V, Porpiglia M, Agresti R, Luini A, Viale G, Cassano E, Peradze N, Toesca A, Massari G, Sacchini V, Munzone E, Leonardi MC, Cattadori F, Di Micco R, Esposito E, Sgarella A, Cattaneo S, Busani M, Dessena M, Bianchi A, Cretella E, Ripoll Orts F, Mueller M, Tinterri C, Chahuan Manzur BJ, Benedetto C, Veronesi P; SOUND Trial Group. Sentinel Lymph Node Biopsy vs No Axillary Surgery in Patients With Small Breast Cancer and Negative Results on Ultrasonography of Axillary Lymph Nodes: The SOUND Randomized Clinical Trial. JAMA Oncol. 2023 Nov 1;9(11):1557-1564. doi: 10.1001/jamaoncol.2023.3759. PMID 37733364
- [Background] Eroglu Z, Krinshpun S, Kalashnikova E, Sudhaman S, Ozturk Topcu T, Nichols M, Martin J, Bui KM, Palsuledesai CC, Malhotra M, Olshan P, Markowitz J, Khushalani NI, Tarhini AA, Messina JL, Aleshin A. Circulating tumor DNA-based molecular residual disease detection for treatment monitoring in advanced melanoma patients. Cancer. 2023 Jun 1;129(11):1723-1734. doi: 10.1002/cncr.34716. Epub 2023 Mar 4. PMID 36869646
- [Background] Bellomo D, Arias-Mejias SM, Ramana C, Heim JB, Quattrocchi E, Sominidi-Damodaran S, Bridges AG, Lehman JS, Hieken TJ, Jakub JW, Pittelkow MR, DiCaudo DJ, Pockaj BA, Sluzevich JC, Cappel MA, Bagaria SP, Perniciaro C, Tjien-Fooh FJ, van Vliet MH, Dwarkasing J, Meves A. Model Combining Tumor Molecular and Clinicopathologic Risk Factors Predicts Sentinel Lymph Node Metastasis in Primary Cutaneous Melanoma. JCO Precis Oncol. 2020;4:319-334. doi: 10.1200/po.19.00206. Epub 2020 Apr 14. PMID 32405608
- [Background] Mulder EEAP, Dwarkasing JT, Tempel D, van der Spek A, Bosman L, Verver D, Mooyaart AL, van der Veldt AAM, Verhoef C, Nijsten TEC, Grunhagen DJ, Hollestein LM. Validation of a clinicopathological and gene expression profile model for sentinel lymph node metastasis in primary cutaneous melanoma. Br J Dermatol. 2021 May;184(5):944-951. doi: 10.1111/bjd.19499. Epub 2020 Nov 2. PMID 32844403
- [Background] Lee RJ, Gremel G, Marshall A, Myers KA, Fisher N, Dunn JA, Dhomen N, Corrie PG, Middleton MR, Lorigan P, Marais R. Circulating tumor DNA predicts survival in patients with resected high-risk stage II/III melanoma. Ann Oncol. 2018 Feb 1;29(2):490-496. doi: 10.1093/annonc/mdx717. PMID 29112704
- [Background] Tie J, Cohen JD, Lahouel K, Lo SN, Wang Y, Kosmider S, Wong R, Shapiro J, Lee M, Harris S, Khattak A, Burge M, Harris M, Lynam J, Nott L, Day F, Hayes T, McLachlan SA, Lee B, Ptak J, Silliman N, Dobbyn L, Popoli M, Hruban R, Lennon AM, Papadopoulos N, Kinzler KW, Vogelstein B, Tomasetti C, Gibbs P; DYNAMIC Investigators. Circulating Tumor DNA Analysis Guiding Adjuvant Therapy in Stage II Colon Cancer. N Engl J Med. 2022 Jun 16;386(24):2261-2272. doi: 10.1056/NEJMoa2200075. Epub 2022 Jun 4. PMID 35657320